CLINICAL TRIAL: NCT03731052
Title: A Double-Blind, Randomized, Multicenter, Vehicle-Controlled, Parallel Group Comparison Study to Determine the Efficacy and Safety of 188-0551 Spray Versus Vehicle Spray in Subjects With Plaque Psoriasis Receiving Up to Four Weeks of Twice-Daily Treatment (Study 307)
Brief Title: Comparison of 188-0551 Spray Versus Vehicle Spray in Subjects With Plaque Psoriasis (307)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 188-0551-307
Record Dates: First submitted 2018-11-02; First posted 2018-11-06 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Plaque Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Drug: 188-0551 Spray (Experimental): 188-0551 Spray applied topically twice daily to psoriatic lesions within the assigned treatment area for up to four (4) weeks
  Interventions: Drug: 188-0551 Spray
- Vehicle Spray (Placebo Comparator): Vehicle Spray applied topically twice daily to psoriatic lesions within the assigned treatment area for up to four (4) weeks
  Interventions: Drug: Vehicle Spray

INTERVENTIONS:
Drug: 188-0551 Spray — Topical Spray containing active drug
  Arms: Drug: 188-0551 Spray
Drug: Vehicle Spray — Topical Spray containing no active drug
  Arms: Vehicle Spray

SUMMARY:
This Phase 3 study (Study 307) has been designed to determine and compare the efficacy and safety of 188-0551 Spray and Vehicle Spray applied twice daily for up to four weeks in subjects with plaque psoriasis. Subjects will be instructed to apply the test article (188-0551 Spray or Vehicle Spray) to all psoriasis plaques within the designated Treatment Area twice daily for four weeks (Study Day 29), unless the investigator verifies the subject's psoriasis has cleared at Day 15, then test article application will be for 2 weeks (Study Day 15).

ELIGIBILITY:
Inclusion Criteria:

1. Subject is male or non-pregnant female and is at least 18 years of age at time of informed consent.
2. Subject has provided written informed consent.
3. Subject has a clinical diagnosis of stable plaque psoriasis involving a minimum of 2% and no more than 10% body surface area (BSA) (excluding the face, scalp, groin, axillae, and other intertriginous areas).
4. Subject has moderate to severe plaque psoriasis.
5. Subject is willing and able to apply the test article as directed, comply with study instructions, and commit to all follow-up visits for the duration of the study.

Females must be post-menopausal , surgically sterile , or use an effective method of birth control. , Women of childbearing potential (WOCBP) must have a negative urine pregnancy test (UPT) at the Baseline Visit.

Exclusion Criteria:

1. Subject has spontaneously improving or rapidly deteriorating plaque psoriasis.
2. Subject has guttate, pustular, erythrodermic, or other non-plaque forms of psoriasis.
3. Subject has palmar/plantar psoriasis.
4. Subject is pregnant, lactating, or is planning to become pregnant during the study.
5. Subject is currently enrolled in an investigational drug or device study.
6. Subject has been previously enrolled in this study and treated with a test article.

Other protocol defined inclusion or exclusion criteria assessed by the study staff may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects rated a treatment success based on the Investigator's Global Assessment (IGA) Success | Day 29
  The primary efficacy endpoint will be the percentage of subjects with IGA treatment success at End of Study (EOS) where EOS is the subject's last completed post-Baseline visit (Day 29).

SECONDARY OUTCOMES:
Percentage of subjects rated a treatment success for each of the clinical signs of psoriasis (scaling, erythema and plaque elevation) | Day 29
  Scaling, erythema and plaque elevation will each be scored on a 5-point scale where 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate, and 4 = severe. These evaluations are an assessment of the overall or "average" degree of each of three key characteristics present within all of the subject's psoriatic lesions in the Treatment Area by the investigator or designee.
Change from Baseline in pruritus score | Day 29
  The proportion of subjects with ≥4 point reduction from Baseline in the Itch Numeric Rating Scale (I-NRS) at Day 29. The I-NRS is based on a 11-point scale where 0 represents "no itching" and 10 represents "worst itch imaginable."
IGA "treatment success" at Day 15 | Day 15
  The proportion of subjects with IGA "treatment success" at Day 15.

CONTACTS AND LOCATIONS:
Overall Officials: Tony Andrasfay, Study Director — Therapeutics, Inc.
Locations (14):
- United States (14):
  - Site 04, Los Angeles, California
  - Site 14, Ocala, Florida
  - Site 01, Macon, Georgia
  - Site 11, Rolling Meadows, Illinois
  - Site 13, Rockville, Maryland
  - Site 10, Clinton Township, Michigan
  - Site 12, Fridley, Minnesota
  - Site 07, Rochester, New York
  - Site 06, High Point, North Carolina
  - Site 05, Norman, Oklahoma
  - Site 03, Philadelphia, Pennsylvania
  - Site 15, Austin, Texas
  - Site 08, San Antonio, Texas
  - Site 02, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No